CLINICAL TRIAL: NCT06946108
Title: Investigation on the Current Situation and Risk Factors Analysis of Exocrine Insufficiency in Chronic Pancreatitis: A Prospective Cohort Investigation Study
Brief Title: Investigation on the Current Situation and Risk Factors Analysis of Exocrine Insufficiency in Chronic Pancreatitis
Acronym: CP-ESRF
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, professor, Changhai Hospital
Other Study IDs: CP-ESRF
Record Dates: First submitted 2025-04-07; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pancreatitis; Pancreatic Exocrine Insufficiency
Keywords: chronic pancreatitis; Pancreatic Exocrine Insufficiency
MeSH Terms: conditions — Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — feces, for the detection of FE-1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- the patients diagnosed with chronic pancreatitis who underwent inpatient care: This hospital-based cohort study enrolled patients diagnosed with chronic pancreatitis (CP) who underwent inpatient care at Shanghai Changhai Hospital (a WHO Collaborating Center for Pancreatology) between June 2022 and September 2024,Voluntary retention of fecal samples for FE-1 detection in CP patients
  Interventions: Diagnostic Test: Detection of Pancreatic Exocrine Function in Patients with Chronic Pancreatitis (CP)

INTERVENTIONS:
Diagnostic Test: Detection of Pancreatic Exocrine Function in Patients with Chronic Pancreatitis (CP) — For CP patients who are hospitalized, they are recruited to voluntarily preserve their feces for the detection of fecal elastase-1 (FE-1) so as to evaluate the pancreatic exocrine function.

SUMMARY:
Pancreatic exocrine insufficiency (PEI) is one of the common complications of chronic pancreatitis (CP). Mild to moderate PEI may present with atypical digestive tract symptoms such as abdominal distension and abdominal pain, while severe PEI can lead to related complications such as foul-smelling stools, steatorrhea, weight loss, and malnutrition. Currently, there is no relevant report on the status quo of PEI in Chinese CP patients. This study aims to analyze the status quo of PEI and related risk factors in Chinese CP patients, with the hope of providing safe and effective intervention and treatment methods to improve the quality of life of patients.

DETAILED DESCRIPTION:
Pancreatic exocrine insufficiency (PEI) is one of the common complications of chronic pancreatitis (CP). Mild to moderate PEI may present with atypical digestive tract symptoms such as abdominal distension and abdominal pain, while severe PEI can lead to related complications such as foul-smelling stools, steatorrhea, weight loss, and malnutrition. Currently, there is no relevant report on the status quo of PEI in Chinese CP patients.This study aims to analyze the current status and related risk factors of PEI in CP patients in China by detecting pancreatic exocrine function with FE-1, in order to provide safe and effective intervention and treatment methods and improve the quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

1. patients who underwent inpatient care at Shanghai Changhai Hospital (a WHO Collaborating Center for Pancreatology) between June 2022 and September 2024.
2. patients diagnosed with chronic pancreatitis (CP)
3. Voluntarily preserve feces for the detection of fecal elastase-1 (FE-1)

Exclusion Criteria:

1. Patients who were diagnosed with pancreatic cancer within 2 years after being diagnosed with chronic pancreatitis (CP)
2. patients with groove pancreatitis,
3. patients with autoimmune pancreatitis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This hospital-based cohort study enrolled patients diagnosed with chronic pancreatitis (CP) who underwent inpatient care at Shanghai Changhai Hospital (a WHO Collaborating Center for Pancreatology) between June 2022 and September 2024
Sampling Method: Non-Probability Sample
Enrollment: 1101 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Detection of Pancreatic Exocrine Function in CP Patients | Day 1
  For CP patients who are hospitalized, they are recruited to voluntarily preserve their feces for the detection of fecal elastase-1 (FE-1) so as to evaluate the pancreatic exocrine function.

SECONDARY OUTCOMES:
The demographic information of the patients | Day 1
  The gender（male/female）, age, height（cm） and weight（kg） upon admission, history of smoking and drinking, family medical history, etc. of the patients with chronic pancreatitis （Only occurrences were recorded as occurring or not occurring）
The information of the patients' natural disease course | Day 1
  The age of onset of chronic pancreatitis (CP), the age of diagnosis, the mode of onset, the type of pancreatic abdominal pain, pancreatic calculi, abnormal blood glucose (impaired fasting glucose, diabetes mellitus), steatorrhea, pseudocyst, common bile duct stricture, pancreatogenic portal hypertension, severe acute pancreatitis (SAP) and the occurrence of other events, etc.（Only occurrences were recorded as occurring or not occurring）
Relevant treatment information for chronic pancreatitis (CP) | Day 1
  Previous treatment methods, the status of pancreatic duct decompression, the morphology of the main pancreatic duct, the in-place condition of the stent after endoscopic surgery, etc.（Only occurrences were recorded as occurring or not occurring）

CONTACTS AND LOCATIONS:
Overall Officials: Liang-hao Hu, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thierens N, Verdonk RC, Lohr JM, van Santvoort HC, Bouwense SA, van Hooft JE. Chronic pancreatitis. Lancet. 2025 Dec 21;404(10471):2605-2618. doi: 10.1016/S0140-6736(24)02187-1. Epub 2024 Dec 5. PMID 39647500
- [Background] Hao L, Wang T, He L, Bi YW, Zhang D, Zeng XP, Xin L, Pan J, Wang D, Ji JT, Du TT, Lin JH, Wang LS, Zou WB, Chen H, Xie T, Guo HL, Li BR, Liao Z, Xu ZL, Li ZS, Hu LH. Risk factor for steatorrhea in pediatric chronic pancreatitis patients. BMC Gastroenterol. 2018 Dec 5;18(1):182. doi: 10.1186/s12876-018-0902-z. PMID 30518343